CLINICAL TRIAL: NCT02965755
Title: Individualized Molecular Analyses Guide Efforts in Breast Cancer - Personalized Molecular Profiling in Cancer Treatment at Johns Hopkins
Brief Title: Personalized Molecular Profiling in Cancer Treatment at Johns Hopkins
Acronym: IMAGE-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Foundation Medicine (Industry); Avon Foundation (Other); Biocept, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J16146; IRB00117742 (Other: JHMIRB)
Record Dates: First submitted 2016-10-18; First posted 2016-11-17 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Breast Cancer; Molecular profiling; Personalized medicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genetic profiling (Other): All participants will undergo genetic profiling. Archival tissue will be requested to undergo routine review for possible treatment recommendations. Blood samples will be obtained to study research correlates (plasma tumor DNA, ptDNA) and tissue comparison.
  Interventions: Other: Treatment recommendation

INTERVENTIONS:
Other: Treatment recommendation — Depending on the results from the participant's archival tissue, a panel of Johns Hopkins investigators will meet to interpret the molecular and genetic profiling results in order to identify any actionable mutations to provide a personalized treatment recommendation for the patient.

SUMMARY:
The goal of this research study is to determine if we can obtain personalized genetic information from a subject's blood sample that is similar to that obtained from a tumor tissue sample, and if we can use that information to make treatment suggestions.

DETAILED DESCRIPTION:
The goal of this research study is to determine if we can obtain personalized genetic information from a subject's blood sample that is similar to that obtained from a tumor tissue sample, and if we can use that information to make treatment suggestions. As tumor samples can be difficult to collect, we hope to be able to collect similar genetic information from blood or urine samples that we find in tumor tissue. Ultimately, we hope to identify genes important to cancer cells that could potentially identify standard-of-care or research-based recommendations for therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 years of age or older
* Metastatic breast cancer and treatment with prior chemotherapy
* Any clinical phenotype (Triple negative, Hormone receptor positive, human epidermal growth factor receptor 2 (HER2)-positive)
* Patient must have received a metastatic tumor biopsy within 3 years prior to the date of the first planned blood sample for the study and have tissue available from this biopsy
* Able to voluntarily provide informed consent

Exclusion Criteria:

* Women who are pregnant or nursing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ability of genetically profiling of ptDNA as assessed by identifying the proportion of genetic alterations in tumor tissue | 1 year
  The proportion of genetic alterations in tumor tissue is detected via genetic profiling of ptDNA when those genetic alterations are present in the tumor at an allelic frequency >10%.
Percentage of patients who cannot have NGS of metastatic site biopsy but have clinically actionable mutations detected via genetic profiling of ptDNA | 1 year
  Percentage of patients for which genetic profiling of ptDNA would be more feasible when a metastatic biopsy cannot be acquired.

SECONDARY OUTCOMES:
Response as assessed by change in ptDNA level up to 2 weeks post-intervention. To determine whether a 10-fold decrease in allelic frequency of a given mutation in ptDNA after initiating new systemic therapy can predict for response to treatment. | 2 weeks
  Change in number-of-folds decrease in allelic frequency of a given mutation in ptDNA 1 or 2 weeks after beginning new systemic therapy.
Response as assessed by Change in Circulating tumor cell (CTC) counts | Change from baseline up to 1 year
  Measure CTC counts at baseline, after 1-2 weeks of therapy, and at each restaging, up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, M.D., Principal Investigator — Johns Hopkins University; Jenna Canzoniero, MD, Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Allegheny Health Network Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.